CLINICAL TRIAL: NCT05208281
Title: Multicenter, Open-Label, Multi-cohort Study to Evaluate Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Drug Product GNR 055 (JSC "GENERIUM", Russia) in Patients With Mucopolysaccharidosis Type II
Brief Title: A Multi-cohort Study of Safety, Efficacy, PK and PD of GNR-055 in Patients With Mucopolysaccharidosis Type II
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDB-MPS-II-III
Record Dates: First submitted 2021-10-14; First posted 2022-01-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mucopolysaccharidosis Type II; Metabolic Diseases
Keywords: Mucopolysaccharidosis type II; Cognitive Dysfunction; Metabolic Diseases; Lysosomal Storage Diseases; Neurocognitive Disorders; Metabolism, Inborn; Genetic Diseases, Inborn; Neurobehavioral Manifestations; Neurologic Manifestations; Genetic Diseases, X-Linked; Hunter syndrome; Iduronate-2-sulfatase; Modified I2S protein; Connective Tissue Diseases; Mental Disorders; Intellectual Disability; Nervous System Diseases; Heredodegenerative Disorders, Nervous System; Cognition Disorders; Mental Retardation, X-Linked
MeSH Terms: conditions — Mucopolysaccharidosis II; Metabolic Diseases; Cognitive Dysfunction; Lysosomal Storage Diseases; Neurocognitive Disorders; Genetic Diseases, Inborn; Neurobehavioral Manifestations; Neurologic Manifestations; Genetic Diseases, X-Linked; Sudden Infant Death; Connective Tissue Diseases; Mental Disorders; Intellectual Disability; Nervous System Diseases; Heredodegenerative Disorders, Nervous System; Cognition Disorders; X-Linked Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adult: GNR-055 (Experimental): GNR-055: 1.0-2.0-3.0 mg/kg
  Interventions: Drug: GNR-055 1.0-2.0-3.0 mg/kg
- Paediatric: GNR-055 2.0 mg/kg (Experimental): GNR-055 2.0 mg/kg
  Interventions: Drug: GNR-055 2.0 mg/kg
- Paediatric: GNR-055 3.0 mg/kg (Experimental): GNR-055 3.0 mg/kg
  Interventions: Drug: GNR-055 3.0 mg/kg

INTERVENTIONS:
Drug: GNR-055 1.0-2.0-3.0 mg/kg — Weekly IV infusion (lyophilized powder) 1.0-2.0-3.0 mg/kg
  Other Names: GNR-055
  Arms: Adult: GNR-055
Drug: GNR-055 2.0 mg/kg — Weekly IV infusion (lyophilized powder) 2.0 mg/kg
  Other Names: GNR-055
  Arms: Paediatric: GNR-055 2.0 mg/kg
Drug: GNR-055 3.0 mg/kg — Weekly IV infusion (lyophilized powder) 3.0 mg/kg
  Other Names: GNR-055
  Arms: Paediatric: GNR-055 3.0 mg/kg

SUMMARY:
This is phase 2/3 study to evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of the investigational product GNR-055 in MPS II (Hunter syndrome) patients of different age groups.

DETAILED DESCRIPTION:
GNR-055 is intended for ERT in patient with Mucopolysaccharidosis type II (MPS II), or Hunter syndrome. MPS II is a recessive X-linked inheritance lysosomal storage disease, which is characterized by a deficiency of the lysosomal enzyme iduronate-2-sulfatase (ID2S), caused by a mutation in the ID2S gene. Enzyme deficiency leads to the accumulation of Glycosaminoglycans (GAG) (mainly of heparan and dermatan sulfates) in lysosomes of almost all types of cells of various tissues and organs. The disease is manifested by growth retardation, damage of many organs and systems, severe deformations of bones and joints, gross facial features, pathology of the respiratory and cardiovascular systems, damage to parenchymal organs (hepatosplenomegaly), and hearing impairment. A severe form of the disease occurs with the involvement of the nervous system in the pathological process, including mental retardation, behavior anomalies, and impaired motor function.

GNR-055 is a recombinant modified ID2S capable to penetrate the blood-brain barrier and thus expected to prevent neurodegenerative consequences and the cognitive deficit and to attain a significant improvement in the life quality and expectancy of patients with MPS II.

Study IDB-MPS-II-III is a multicenter, open-label, multi-cohort study to assess safety, PK and PD, and efficacy of GNR-055 in patients of different age groups with MPS II (Hunter syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent;
* Verified diagnosis of MPS II (Hunter syndrome);
* Naïve patients or patients who have received standard ERT whit idursulfase products;
* No contraindications for lumbar puncture as judged by the Investigator;
* Willingness and ability to follow study procedures.

Exclusion Criteria:

* Clinically pronounced hypersensitivity to ID2S or any other component of the drug product;
* History of hematopoietic stem cell transplantation (HSCT) or bone marrow transplantation;
* Implanted or external non-removable metal devices, a cardiac pacemaker, or other objects sensitive to the magnetic field that may pose a danger to both the wearer and the correct operation of magnetic resonance imaging (MRI) equipment;
* Concomitant diseases and conditions that, in the Investigator's opinion, can put at risk the patient's safety during his/her participation in the study, or which will influence the safety data analysis in case of the disease/condition exacerbation during the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events (AEs) and Serious Adverse Events (SAEs) | Baseline to Week 56
  Safety assessment will be performed based on the subjective complaints, physical examination, assessment of vital signs, laboratory tests, and 12-lead ECG; Incidence of allergic and infusion-related reactions; Incidence of Anti-Drug Antibodies (ADAs) against GNR-055 and their neutralizing activity.
Urine GAG excretion | Baseline to Week 4, 8, 10, 26, and 52
  Changes in levels of urine GAG excretion after multiple-dose administration of GNR-055

SECONDARY OUTCOMES:
Serum concentration of the GNR-055 | Week 52
  Assessment of the serum concentration of GNR-055 and calculation of Cmax, AUC, T1/2, Cl et other parameters after multiple-dose administration
GAG level in CerebroSpinal Fluid (CSF) | Baseline to Week 6, 10, 26, and 52
  Changes in levels of CSF GAG after multiple-dose administration of GNR-055
Serum GAG level | Baseline to Week 4, 8, 10, 26, and 52
  Changes in levels of serum GAG after multiple-dose administration of GNR-055
Large joint range of motion | Week 8, 10, 26, and 52
  Changes over time in the large joint range of motion after multiple-dose administration of GNR-055
Liver and spleen volumes (MRI) | Baseline to Week 8, 10, 26, and 52
  Changes over time in liver and spleen volume according to ultrasound/MRI after multiple-dose administration of GNR-055
6-minute walk test | Baseline to Week 8, 10, 26, and 52
  Changes over time in the results of the 6-minute walk test after multiple-dose administration of GNR-055
Left ventricular mass by EchoCG | Baseline to Week 8, 10, 26, and 52
  Changes over time in the left ventricular mass according to Echocardiography (Echo-CG) after multiple-dose administration of GNR-055
Lung Forced Vital Capacity (FVC) | Baseline to Week 8, Week 26, and Week 52
  Changes over time in FVC according to spirometry after multiple-dose administration of GNR-055
Neurocognitive functions assessment | Baseline to Week 12, 26, and 52
  Changes over time in neurocognitive functions after multiple-dose administration of GNR-055
Brain white/gray matter structures (MRI) | Baseline to Week 26, and 52
  Changes over time in the quantitative MRI brain structure parameters after multiple-dose administration of GNR-055
Serum neuromarkers | Baseline to Week 24, and 52
  Changes in levels of serum neuromarkers after multiple-dose administration of GNR-055
CSF neuromarkers | Baseline to Week 24, and 52
  Changes in levels of CSF neuromarkers after multiple-dose administration of GNR-055

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, MSc, Study Director — AO GENERIUM
Locations (5):
- Russia (5):
  - Federal State-Funded Healthcare Institution Central Clinical Hospital of the Russian Academy of Sciences (Research Institute of Pediatrics and Child Health Protection of the Central Clinical Hospital of the Russian Academy of Sciences), Moscow
  - Federal State Budgetary Educational Institution of Higher Education "St. Petersburg State Pediatric Medical University" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - V.I. Vernadsky Crimean Federal University, Simferopol
  - State Budgetary Healthcare Institution Republican Medical Genetic Center, Ufa
  - State Autonomous Healthcare Institution of the Sverdlovsk Region Regional Children's Clinical Hospital, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No